CLINICAL TRIAL: NCT06252129
Title: Maximizing Lymph Node Dissection on Fresh and Fixed Lung Cancer Resection Specimens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Paula Antonia Ugalde Figueroa, Associate Surgeon, Division of Thoracic Surgery, Principal Investigator., Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DFCI IRB protocol #23-576
Record Dates: First submitted 2023-12-21; First posted 2024-02-09 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer; Lymph Node Metastasis; Pathologic Processes
Keywords: NSCLC; Lymph node dissection; Lung cancer staging
MeSH Terms: conditions — Lung Neoplasms; Lymphatic Metastasis; Pathologic Processes | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Interventional group (Experimental): subjects who are being consented to this study and undergoing lymph node dissection as outlined in this protocol
- Concurrent non-interventional group (No Intervention)
- Retrospective cohort from 2021-2020 (Other)
  Interventions: Other: Control group

INTERVENTIONS:
Other: Subjects undergoing a lung specimen lymph node dissection — A lobectomy specimen's resection will undergo systematic lymph node dissection either by the patient's treating thoracic surgeon and/or by a member of the pathology team.
  The protocol for a standardized lymph node dissection consists of a series of blunt peribronchial dissections starting from the hilum to the periphery, with particular attention to points of airway bifurcation where intrapulmonary lymph nodes aggregate. By emphasizing the intrapulmonary lymph node map and a standardized dissection, the team will remove more lymph nodes from the lobectomy specimen, resulting in an accurate N staging.
Other: Control group — Control group
  Arms: Retrospective cohort from 2021-2020

SUMMARY:
Lung cancer patients undergoing upfront surgery, highly benefit from a systematic lymph node dissection in the mediastinum and in the surgical specimens. The latter is performed by the pathologist. Developing a standardized technique to dissect the lobectomy specimen has the potential of maximizing the retrieval of all N1 stations lymph nodes. The investigators believe that the adoption of such technique will improve lung cancer staging and identify a higher number of patients that qualify for adjuvant therapies.

DETAILED DESCRIPTION:
Anatomic lung resection with systematic mediastinal lymph node dissection is the standard of care for patients with clinical stage I or II non-small cell lung cancer (NSCLC). While the best type of resection may sometimes be debated, it is clear that mediastinal, hilar, and lobar lymph nodes (LNs) should be routinely retrieved to achieve a complete lung cancer resection. According to major international guidelines, at least 3 hilar/intrapulmonary stations and 3 mediastinal stations should be assessed during resection. Although there is still a debate over whether the ideal number of LN stations sampled or the total number of LNs removed per station provides a better analysis, radical systematic LN dissection seems to offer the best oncological outcomes. In fact, in patients with tumors ≤4 cm in diameter completely resected, the quality of the mediastinal lymph node dissection and the thoroughness of the examination of the surgical specimen will select candidates for adjuvant treatment and define oncologic prognosis. The consequences of an incorrect lymph node classification can be substantial: while patients with N0 NSCLC have approximately 75% 5-year overall survival (OS), patients with NSCLC classified as N1 have a 5-year OS of 49%, and patients with NSCLC classified as N2 a 5-year OS of 36%. Therefore, the burden of determining the correct prognosis lies on the surgeon to perform a rigorous and thorough oncological resection, and on the pathologist to fully assess enough intrapulmonary LNs. Inaccuracy by either specialist leads to pathologic understage and suboptimal clinical management, which will lead to poor patient outcomes.

Developing a standardized technique to dissect the lobectomy specimen has the potential of maximizing the retrieval of all N1 stations lymph nodes. The investigators believe that the adoption of such technique will improve lung cancer staging and identify a higher number of patients that qualify for adjuvant therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a lung nodule or mass who are eligible to undergo a lobectomy.
2. Subject without any metastasis present.
3. Subjects who have peripheral lung nodule location
4. Subjects must be 18 years of age or older.

Exclusion Criteria:

1. Subjects who received preoperative chemotherapy or radiotherapy.
2. Subjects who have a lung nodule located in a central location. Central tumors are defined by those infiltrating the lobar airway.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of lymph nodes sampled | 2 weeks
  To compare the number of stations and lymph nodes sampled when adopting a standardized technique compared to the conventional (prior) technique.
Nodal upstage rate | 2 weeks
  Determine the number of cases upstaged to N1 with the intrapulmonary lymph node dissection compared to the conventional technique.

SECONDARY OUTCOMES:
3y RFS | 3 years
  Three years recurrence-free survival rate of patients undergoing standardize dissection versus conventional technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Womens Hospital, Boston, Massachusetts, United States